CLINICAL TRIAL: NCT06947343
Title: Effect of Action Observation Therapy in Comparison to Motor Relearning Program on Balance and Mobility Among Subacute Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/66
Record Dates: First submitted 2025-04-20; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Subacute Stroke; Cerebral Stroke; Cerebrovascular Stroke; Posture; Functional Performance
Keywords: Action observation therapy; Motor relearning program
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Action Observation Therapy GROUP (Experimental): functional AOT with visual feedback and physcial training after watching a video 30mins session, 3times/week total 8weeks 3mins for observation phase, 2min for action execution stage 1, sitting position (static and dynamic balance) exercies for trunk flexion, upper and lower trunk rotation multidirectional reaching to pickup any object from different directions,foward,lateral and diagnol reaching stage 2, sit to stand and stand to sit from sitting to standing, trunk flexed, hips and knees 90 degree flexed, feet behind knee, 15cm apart, then standing, trunk extension hips knees extend feet apart and viceversa 4phases of sit to stand, seat off, standing, seat on, sitting in sitting position dorsiflexion training, flexion extension training knee joint the right hand touches the left foot and viceversa
  Interventions: Procedure: ACTION OBSERVATION THERAPY
- Motor Relearning Program Group (Experimental): Motor relearning program based on task oriented training 30mins, 3times/week total 8weeks stage 1, balanced sitting exercises for trunk flexion and rotation, feet and knees 15cm apart multidirectional reaching while seated forward, lateral and diagnol reaching to pick up any thing from different directions butt walking scooting on bed stage 2, standing up and sitting down transition from a seated position on a firm flat surface with no armrests to standing with an upright posture, upper body vertical and feet placed backward followed by sitting down by flexing hips,knees and ankle prerequisited of sit to stand, 4phases in sitting dorsiflexion training, flexion extension training of knee joint right hand touch to left foot and viceversa picking up objects from floor stage3, balanced standing weight shifting head and trunk movemnts while standing with feetapart standing unsupported with eyes closed multidirectional reaching, forward, bakcward, lateral and diagonal
  Interventions: Procedure: MOTOR RELEARNING PROGRAM

INTERVENTIONS:
Procedure: ACTION OBSERVATION THERAPY — functional AOT with visual feedback and physical training after watching a video 30mins session, 3times/week total 8weeks 3mins for observation phase, 2min for action execution Stage 1, sitting position (static and dynamic balance) exercises for trunk flexion, upper and lower trunk rotation multidirectional reaching to pick up any object from different directions, forward, lateral, and diagonal reaching Stage 2, sit to stand and stand to sit from sitting to standing, trunk flexed, hips and knees 90 degree flexed, feet behind knee, 15cm apart, then standing, trunk extension hips knees extend feet apart and vice vers 4phases of sit to stand, seat off, standing, seat on, sitting in sitting position dorsiflexion training, flexion extension training knee joint the right hand touches the left foot and viceversa pick up an object from floor stage3, standing balance weight shifting, front, back, sideways, left and right head and trunk movements in different directions while standing
  Arms: Action Observation Therapy GROUP
Procedure: MOTOR RELEARNING PROGRAM — Motor relearning program, interventional group B, based on task-oriented training 30mins, 3times/week total 8weeks stage 1, balanced sitting exercises for trunk flexion and rotation, feet and knees 15cm apart multidirectional reaching while seated forward, lateral and diagonal reaching to pick up any thing from different directions butt walking scooting on bed stage 2, standing up and sitting down transition from a seated position on a firm flat surface with no armrests to standing with an upright posture, upper body vertical and feet placed backward followed by sitting down by flexing hips,knees and ankle prerequisited of sit to stand, 4phases in sitting dorsiflexion training, flexion extension training of knee joint right hand touch to left foot and viceversa picking up objects from floor stage3, balanced standing weight shifting head and trunk movemnts while standing with feetapart standing unsupported with eyes closed multidirectional reaching
  Arms: Motor Relearning Program Group

SUMMARY:
This study is a randomized controlled trial. The purpose of this study is to determine the effect of Action Observation Therapy in Comparison to a Motor Relearning Program on Balance and Mobility among subacute stroke patients.

DETAILED DESCRIPTION:
Action observation therapy has proven its positive effects in improving functional performance in stroke patients compared to other neurological and musculoskeletal conditions motor relearning program is also very effective in improving functional performance in stroke patients but previous studies have shown individual effects of AOT and MRP but there is no comparison of AOT with MRP on balance and mobility.

as a result, this study aims to contribute new data to the sparse literature on subacute stroke patients.

The research finidings could provide valuable insights into potential benefits, encouraging evidence-based practices.

ELIGIBILITY:
Inclusion Criteria:

* Both genders, male and female
* Ischemic stroke patients
* Age 45 years and above
* MMSE>24
* Able to stand independently for 1 minute
* Patient can maintain starting sitting static position for 10 seconds without arm rest

Exclusion Criteria:

* Any other neurological disorder
* Orthopedic conditions(fracture) affecting balance and mobility
* Visual or auditory impairments

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Balance | 8 weeks
  Berg Balance Scale will be used to assess balance
anticipatory balance | 8 weeks
  Modified functional reach test will be used
Mobility | 8 weeks
  The timed up and go test will be used

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan